CLINICAL TRIAL: NCT01373476
Title: Multicentre,Randomized,Double-blind, Multiple-dose, Placebo-controlled, Parallel-Group Trial of Qideng Mingmu Capsule in The Treatment of Diabetic Retinopathy With Blood Stasis Syndrome and Deficiency of Qi-Yin Syndrome
Brief Title: Multicentre, Randomized, Controlled Trial of Qideng Mingmu Capsule in The Treatment of Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Chongqing Taiji Group of Fuling pharmaceutical Co., LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2008L11200
Record Dates: First submitted 2011-04-26; First posted 2011-06-15 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Diabetic Retinopathy; Diabetic Eye Problems; Retinal Disorders
Keywords: Diabetic Retinopathy; Traditional Chinese medicine; Diabetic Eye Problems; Retinal Disorders
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qideng Mingmu capsule (Experimental): High dosage group,Middle dosage group,Low dosage group.
  Interventions: Drug: Qideng Mingmu capsule
- Placebo (Placebo Comparator): Placebo group
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Qideng Mingmu capsule — High dosage group (4 Qideng Mingmu capsules each time): 4#, po, tid,24 weeks; Middle dosage group (2 Qideng Mingmu capsules plus 2 placebos each time):4#, po, tid,24 weeks;Low dosage group (1 Qideng Mingmu capsule plus 2 placebos each time):3#, po, tid,24 weeks.
  Arms: Qideng Mingmu capsule
Drug: Placebo Comparator — Placebo group (4 placebos each time):4#, po, tid,24 weeks.
  Arms: Placebo

SUMMARY:
Objectives of study: To preliminarily evaluate the efficacy and safety of Qideng Mingmu Capsule in the treatment of patients with diabetic retinopathy (deficiency of Qi-Yin syndrome, blood stasis syndrome), to discuss the appropriate dose and period of treatment.

DETAILED DESCRIPTION:
The efficacy of Qideng Mingmu capsule is to nourish qi-yin and promote blood circulation. It is used in patients with diabetic retinopathy who are differentiated as deficiency of Qi-Yin syndrome and blood stasis syndrome in traditional Chinese medicine(TCM).The manifestation of diabetic retinopathy(DR) mainly includes dim and dry eyes,shortness of breathe, fundus hemorrhage,etc.The experimental research indicated that the Qideng Mingmu capsule could improve the GK rats' quality of life,through reducing vascular endothelial growth factor(VEGF) level in vitreous of GK rats and inhibiting the expression of protein kinase C(PKC),therefore is capillary protective agent against retinal impairment in GK rat.The toxicology test has proved that the clinical dosage of Qideng Mingmu capsule is safe.Both acute and long-term toxicity tests has showed no toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-proliferative diabetic retinopathy(NPDR)，differentiated as deficiency of Qi-Yin syndrome or blood stasis syndrome in traditional Chinese medicine(TCM).
* best-corrected ETDRS visual acuity in study eye≥15 letters,or about 0.16(20/125) by the decimal point method.
* Age between 30 and 70 years old.
* Able and willing to give informed consent
* Keep the level of blood sugar steady during the last three months before randomization, meanwhile the glucose lowering therapy could be predicted without any change during this study.
* Eligible patients are with moderate and severe diabetic retinopathy primarily, mild of whom are controlled within 15%.
* All procedures from participance in the study voluntarily, signature on the Informed Consent Form (ICF) and acceptance of treatment are according to GCP guidelines.

Exclusion Criteria:

* Patients with ineffective blood sugar control (HbAlc>9%) or without usage of fundamental antidiabetic drugs such as biguanides, sulfonylureas (SUs), insulin and thiazolidinediones (TZDs).
* Patients who have had intraocular surgery like retina photocoagulation within 6 month; or are appropriate for laser photocoagulation currently, on the condition that more than two quadrants have extensive non-perfusion areas.
* Patients with other ophthalmological combined diseases like glaucoma, cataract that have effected the check of eyeground deeply, non-diabetic retinopathy, uveitis, retinal detachment, diseases of optic nerve, high myopia with eyeground pathological changes,etc.
* Patients with severe cardiovascular diseases, functional disorders of liver and kidneys, diseases of the haematopoietic system (bone marrow hypoplasia, leucopenia, anemia, etc.), severely abnormal electrocardiogram (ECG), ALT>2 *ULN, Cr >1.5*ULN and psychopaths.-Patients with diabetic nephropathy (DN) in the stage of azotemia or uremia.
* Pregnant women or trying to conceive or in lactation; patients with allergic constitution.
* Patients who have participated in other clinical trials in recent one month.
* Patients who have used the drugs in the treatment of diabetic retinopathy (calcium dobesilate, Difrarel, capsule of Xueshuantong, ginkgo biloba extract, Qiming granula, etc.) in past two weeks.
* Patients with SBP>160mmHg or DBP﹥100mmHg.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Ocular fundus | Change from Baseline in Ocular fundus which is to be examined by color fundus image at 6 months

SECONDARY OUTCOMES:
Fundus fluorescein angiography (FFA) | at baseline phase and 24 weeks after randomization
  Fundus fluorescein angiography (FFA) is to be tested at baseline phase and 12, 24 weeks after randomization, which will provide details of retinal circulation time(retinal arterial stage, capillary transition stage and venous stage included),non-perfusion areas in capillary of the retina(location and range noted),and leakage from the retinal vessels(location and range noted).
best-corrected ETDRS visual acuity | at baseline phase and every four weeks after randomization.
  best-corrected ETDRS visual acuity will be captured at baseline phase and every four weeks after randomization.
Traditional Chinese medical (TCM) syndrome scores | at baseline phase and every four weeks after randomization.
  Traditional Chinese medical (TCM) syndrome scores will be collected at baseline phase and every four weeks after randomization.
the observation of Ocular fundus | at baseline phase and 12, 24 weeks after randomization
  Ocular fundus is to be examined by color fundus image at baseline phase and 12, 24 weeks after randomization, reflecting the abnormality of intraretinal microvasculature.
Optic coherence tomography (OCT) | at baseline phase and 12, 24 weeks after randomization
  Optic coherence tomography (OCT) is to be tested at baseline phase and 12, 24 weeks after randomization, indicating the degree of macular edema.

CONTACTS AND LOCATIONS:
Overall Officials: Fuwen Zhang, Ph.D, Study Director — Chengdu University of Traditional Chinese Medicine
Locations (8):
- China (8):
  - Beijing Tongren Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Daping Hospital of Third Military Medical University, Chongqing, Chongqing Municipality
  - Guangdong Province Traditional Medical Hospital, Guangzhou, Guangdong
  - The first affiliated hospital of Hunan University of TCM, Changsha, Hunan
  - Jiangsu Province Traditional Medical Hospital,, Nanjing, Jiangsu
  - Affiliated Hospital of Chengdu University of TCM, Chengdu, Sichuan
  - West China Hospital, Chengdu, Sichuan
  - The first affiliated hospital of Guangzhou university of TCM, Guangzhou